CLINICAL TRIAL: NCT06436872
Title: The Effect of Informatıon Provıded to the Relatıves of Patıents Undergoıng Open Heart Surgery on the Qualıty of Lıfe and Caregıver Burden.
Brief Title: The Effect of Informing the Relatives of Patients Undergoing Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Esra Akdeniz, BSN Nurse, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GOBAEK-2022/206
Record Dates: First submitted 2024-03-19; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Open Heart Surgery; Life Quality; Caregiver Burden
Keywords: open heart surgery; life quality; caregiver burden; nursing information
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysed by a independent researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Caregivers in the study group were given 45 minutes of training and a booklet in line with the training booklet prepared according to daily life activities aimed at improving the patient's quality of life and reducing the caregiver's care burden. The caregivers in the study group were given the researcher's contact number and were able to reach the researcher whenever they needed.
  Interventions: Other: informing patients with using a booklet
- Control Group (No Intervention): Patients in the control group underwent standard procedure; No information, training booklet or contact number was provided. The Caregiver Information Form was administered by the researcher in a face-to-face meeting with the caregiver. The Patient Introduction Form was filled out by the researcher from the patients' files. Multidimensional Quality of Life Scale was administered by the researcher. The Caregiving Burden Scale was introduced to the caregiver by the researcher and filled in by the caregiver himself. The Caregiver Tracking Form, prepared to track the patient and the caregiver, was applied to the caregiver by the researcher in order to determine the caregiver's zero point.

INTERVENTIONS:
Other: informing patients with using a booklet — The intervention group was informed before discharge and was given an information booklet. A phone number was given so that the researcher could contact the nurse. In the 4th week, 8th week and 12th week, information was given according to the information needs of the patient and caregiver.
  Arms: intervention group

SUMMARY:
The goal of this type of study clinical trial is to determine the effect of informing the relatives of patients undergoing open heart surgery on the patients; quality of life and caregiver burden.The main question it aims to answer are:

H1: Informing caregivers of patients undergoing open heart surgery improves the quality of life of patients.

H2: Informing caregivers of patients undergoing open heart surgery reduces caregiver burden.Relatives of patients who have undergone open heart surgery will be informed about home care before discharge. The researcher will compare the study group with the control group to see if the information given to the caregiver makes a difference on the patient's quality of life.

DETAILED DESCRIPTION:
In the study, patients were assigned to the study and control groups via the randomizer.org website.

The Caregiver Information Form was administered by the nurse researcher in a face-to-face meeting with the caregiver. The Patient Introduction Form was filled out by the researcher from the patients'; files. The Multidimensional Quality of Life Scale was administered by the researcher through a face-to-face interview with the patient. The Caregiving Burden Scale was introduced to the caregiver by the researcher and filled in by the caregiver himself. The Caregiver Tracking Form, prepared to track the patient and the caregiver, was applied to the caregiver by the researcher in order to determine the caregivers zero point. The first data collection was carried out 48 hours after the patient was admitted to the service and before information was given. Caregivers in the study group were given 45 minutes of training and a booklet in line with the training booklet prepared according to daily life activities aimed at improving the patients quality of life and reducing the caregiver's care burden. The caregivers in the study group were given the researcher's contact number and were able to reach the researcher whenever they needed.

Patients in the control group underwent standard procedure; No information, training booklet or contact number was provided. The Caregiver Information Form was administered by the researcher in a face-to-face meeting with the caregiver. The Patient Introduction Form was filled out by the researcher from the patients'; files. Multidimensional Quality of Life Scale was administered by the researcher. The Caregiving Burden Scale was introduced to the caregiver by the researcher and filled in by the caregiver himself. The Caregiver Tracking Form, prepared to track the patient and the caregiver, was applied to the caregiver by the researcher in order to determine the caregiver's zero point. Initial data were collected between 48 hours after the patient was admitted to the ward and before discharge.

Caregiving burden scale and multidimensional quality of life form were applied to both groups at the 4th week, 8th week and 12th week. Patients in the intervention group were informed again according to their needs.

ELIGIBILITY:
Inclusion Criteria for patients:

* Over 65 years of age,
* Does not have any psychological problems and can communicate in Turkish
* Literate,
* Having undergone open heart surgery for the first time
* After being taken to the Cardiovascular Surgery Service, they are stable after completing the 48-hour critical period,
* Elderly individuals who agreed to participate in the research constituted the patient sample of the study.

Inclusion Criteria for caregivers

* The person who is primarily responsible for the patient care and will accompany the patient for 12 weeks, Caregivers,
* Between the ages of 18-65,
* Does not have any psychological problems and can communicate in Turkish,
* The caregiver sample was created by caregiver individuals who agreed to participate in the research.

Exclusion Criteria for patients:

* Those with neurological or metabolic diseases that may cause functional disability
* Previously had open heart surgery
* Patients with mental and cognitive dysfunction
* Patients who did not attend at least one of the post-surgical evaluations for any reason were excluded from the sample.

Exclusion Criteria for caregivers

* Those with neurological or metabolic diseases that may cause functional disability
* Transferring the patient care to someone else during the 12-week working period,
* Caregivers who did not attend at least one of the post-surgical evaluations for any reason were excluded from the sample.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Multidimensional quality of life scale | 12 weeks
  The multidimensional quality of life scale, which is psychometrically strong, short, easy to apply and suitable for patients diagnosed with Cardiovascular Disease, is a tool developed by Avis et al. for the purpose of multidimensional measurement of HRQoL and whose Turkish validity and reliability was obtained by Demir. The total score of the scale varies between 35-245.
Caregiver burden scale | 12 weeks
  It was developed by Zarit, Reever and Bach-Peterson in 1980 to evaluate the stress experienced by caregivers of individuals in need of care. The evaluation of the scale is made based on the total score, and a minimum of 0 and a maximum of 88 points can be obtained from the scale. . 0-20 points obtained from the scale are classified as "little/no burden", 21-40 points as "moderate burden", 41-60 points as "severe burden" and 61-88 points as "extreme burden". A high scale score indicates that the distress experienced is high.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Akdeniz, BSN, Principal Investigator — Trakya Üniversite
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No